CLINICAL TRIAL: NCT07106034
Title: Clinical Study of Second-Line Standard Therapy Combined With Ongericimab and Toripalimab in Patients With MSS/pMMR Colorectal Cancer Following First-Line Treatment Failure
Brief Title: Standard Second-line Therapy With ONgericimab and TOripalimab in pMMR/MSS Colorectal Cancer: a Single-arm Phase II Trial
Acronym: ONTOP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONTOP
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Advanced Colorectal Cancer
Keywords: Toripalimab; Ongericimab; colorectal cancer; pMMR/MSS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second-line standard treatment combined with Ongericimab and toripalimab. (Experimental): If first line treatment with irinotecan-containing regimen:
  Ongrezicimab + Toripalimab + Bevacizumab + FOLFOX, Q2W
  If first line treatment with oxaliplatin-containing regimen:
  Ongrezicimab + Toripalimab + Bevacizumab + FOLFIRI, Q2W
  In addition, the period of 21 days after the first administration is defined as the DLT observation period.
  Interventions: Drug: Ongericimab + Toripalimab + Bevacizumab + FOLFOX; Drug: Ongericimab + Toripalimab + Bevacizumab + FOLFIRI

INTERVENTIONS:
Drug: Ongericimab + Toripalimab + Bevacizumab + FOLFOX — Ongericimab, Toripalimab, Bevacizumab, Oxaliplatin, Calcium folinate, 5-FU, Q2W
Drug: Ongericimab + Toripalimab + Bevacizumab + FOLFIRI — Ongericimab, Toripalimab, Bevacizumab, Irinotecan, Calcium folinate, 5-FU, Q2W

SUMMARY:
The ONTOP study is a prospective, single-arm, open-label phase II clinical trial. A total of 32 patients with advanced MSS/pMMR colorectal cancer who have failed first-line treatment will receive second-line standard treatment combined with Ongericimab and toripalimab. Among them, patients who received irinotecan-containing treatment in the first line will be administered the regimen of Ongericimab + toripalimab + bevacizumab + FOLFOX. Patients who received oxaliplatin-containing treatment in the first line will be administered the regimen of Ongericimab + toripalimab + bevacizumab + FOLFIRI. Treatment will continue until disease progression, initiation of new anti-tumor treatment, active request of the subject, or determination by the investigator that study drug administration needs to be terminated. The primary study endpoint is the objective response rate (ORR), and the secondary study endpoints include duration of response (DoR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and safety, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-75 years (inclusive of 18 and 75 years) at the time of signing the informed consent, regardless of gender.
2. Histologically confirmed MSS/pMMR colorectal or rectal cancer, who have progressed on first-line fluoropyrimidine - based combination therapy (including progression during maintenance therapy). If FOLFOXIRI was received in the first - line, screening is not allowed; if progression occurred during neoadjuvant/adjuvant therapy or within 6 months after the last dose, it is considered first-line treatment failure, and the patient is eligible for enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Predicted survival ≥ 12 weeks.
5. At least 1 measurable lesion according to RECIST 1.1 evaluation criteria.
6. Adequate organ function；
7. Female or male subjects with childbearing potential must agree to have no childbearing plans within 6 months after the end of the last dose during the study period and be willing to take highly effective contraceptive measures together with their partners. For female subjects with childbearing potential, the serum pregnancy test must be negative within 7 days before the first dose, and they must be non - lactating.
8. Be able to provide a signed informed consent form, including complying with the requirements and restrictions listed in the Informed Consent Form (ICF) and this protocol.

Exclusion Criteria:

1. Presence of leptomeningeal metastasis; presence of active brain metastasis, defined as untreated and/or having clinical symptoms, or requiring glucocorticoids or antiepileptic drugs to control related symptoms. For those who have received local treatments such as surgery or radiotherapy, if the screening - period imaging assessment shows no evidence of progression for at least four weeks and symptoms disappear (except for residual signs or symptoms related to brain metastasis), no glucocorticoid treatment is needed for at least 2 weeks, and the acute toxicities related to previous treatments have recovered, enrollment is allowed.
2. Presence of pleural effusion, peritoneal effusion, or pericardial effusion with clinical symptoms or requiring repeated management (such as puncture or drainage).
3. History of immunodeficiency disorders, including positive detection of human immunodeficiency virus (HIV), or known allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
4. History of severe cardiovascular diseases, including but not limited to: myocardial infarction within 6 months before the first study drug administration, severe/unstable angina pectoris, congestive heart failure (NYHA heart function class ≥2), severe supraventricular or ventricular arrhythmia, aortic aneurysm requiring surgical repair, any arterial thromboembolic event, grade 3 or above venous thromboembolic event, transient ischemic attack, cerebrovascular accident.
5. Presence of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months before the first drug administration.
6. Severe infection within 28 days before the first study drug administration (CTCAE 5.0 ≥ grade 2), such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; active infection requiring intravenous anti-infection treatment or unexplained fever > 38.5°C within 2 weeks before the first study drug administration (judged by the researcher; fever caused by the tumor in the subject can be enrolled).
7. Presence of active tuberculosis, hepatitis B (hepatitis B surface antigen [HBsAg] positive and HBV DNA higher than the lower limit of detection of the research center), hepatitis C (HCV Ab positive and HCV RNA higher than the lower limit of detection of the research center).
8. History of another primary malignant tumor, except for those who have received radical treatment before the first administration of the study intervention, have no known active disease (for more than 5 years), and have a low potential recurrence risk (such as skin basal cell carcinoma and cutaneous squamous cell carcinoma that have received curative treatment).
9. The following situations do not allow screening:

   1. Screening period imaging shows that the tumor encircles important blood vessels or has obvious necrosis and cavity, and the researcher deems it may cause bleeding risk;
   2. Clinical signs or symptoms of intestinal obstruction and/or gastrointestinal obstruction within 6 months before the first drug administration, including incomplete obstruction related to the underlying disease;
   3. Presence of severe, unhealed, or ruptured wounds, active ulcers, or untreated fractures;
   4. Clinically significant hemoptysis (≥1/2 tea spoon) or tumor bleeding for any reason within 1 month before the first drug administration;
   5. Presence of poorly controlled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure > 100 mmHg), or history of hypertensive emergency or hypertensive encephalopathy;
   6. Other situations judged by the researcher as unsuitable for receiving oral chemotherapy.
10. Previous antineoplastic treatment toxicity has not recovered to grade 1 specified in CTCAE 5.0 or the level specified in the enrollment/exclusion criteria. Except for the following situations: if the researcher judges that the related toxicity is well-controlled and does not affect the safety and compliance of the subject using the study drug, screening is allowed.
11. Previous occurrence of drug-related adverse events leading to permanent drug discontinuation during treatment with bevacizumab and similar drugs.
12. Received the following drugs or treatments before the first drug administration:

    1. Received chemotherapy, immunotherapy, radiotherapy, and other antineoplastic treatments within 21 days before the first drug administration; received oral fluoropyrimidines, small molecule targeted drugs, antineoplastic vaccines, and intravesical administration (such as BCG for bladder cancer) within 14 days before the first drug administration; started palliative radiotherapy for painful lesions within 7 days before the first drug administration;
    2. Underwent needle biopsy or other minor surgeries (excluding placement of vascular access devices) within 28 days before the first drug administration;
    3. Subjects who used systemic corticosteroids (≥10 mg prednisone equivalent per day) or other immunosuppressants for systemic treatment within 2 weeks before the first drug administration; inhalation or local use of corticosteroids or preventive medication (such as for infusion reaction/hypersensitivity reaction) is allowed;
    4. Received any live vaccine or attenuated vaccine within 28 days before the first drug administration, or need to receive live vaccines during the study period.
13. Used antiplatelet therapy or anticoagulant therapy for therapeutic purposes within 10 days before the first drug administration.
14. Pregnant or lactating women.
15. Presence of other severe physical or mental diseases or abnormal laboratory examinations, which may increase the risk of participating in the study, affect treatment compliance, or interfere with the study results, and are judged by the researcher as unsuitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | Two years
  overall response rate

SECONDARY OUTCOMES:
Disease control rates | Two years
  Disease control rates
Duration of Response | Two years
  Duration of Response
progression-free survival | Two years
  progression-free survival
overall survival | Two years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided